CLINICAL TRIAL: NCT02897986
Title: Study of a Propranolol (HEMANGIOL®) and Oral Metronomic Vinorelbine (NAVELBINE®) Combination for Children and Teenagers With Refractory/Relapsing Solid Tumors
Acronym: PROVIN
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-06
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms | interventions — Vinorelbine

ARMS (1):
- patients with refractory/relapsing solid tumors (Experimental)
  Interventions: Drug: administration of a propranolol (HEMANGIOL®) and oral metronomic vinorelbine (NAVELBINE®) combination

INTERVENTIONS:
Drug: administration of a propranolol (HEMANGIOL®) and oral metronomic vinorelbine (NAVELBINE®) combination

SUMMARY:
Cancer remains the first cause of death due to disease in children and adolescents despite important progress and 70% of the survivors present sequelae. It is therefore mandatory to generate new and preferably less toxic treatment strategies relying on new anticancer agents, and/or new combinations or schedules of administered compounds.

Metronomic chemotherapy (MC) consists in administrating low doses of anticancer agents on a daily/weekly basis. MC has been showed to be a safe and effective way to administer chemotherapy to obtain anti-cancer effects through anti-angiogenic and pro-imune effects.

Drug repositioning consist in using non-anticancer drug for which anti-cancer properties have been unveiled. Propranolol is a non selective beta-blocker initially used to treat hypertension but recently its anticancer properties have been discovered. The place of Betablockers as anticancer agents is supported by both preclinical and epidemiologic data. The investigators have showed that the use of betablockers could sensitize breast cancer, angiosarcoma and neuroblastoma to chemotherapy in vitro and in vivo at least in part via an anti-angiogenic mechanism. There are currently 12 clinical trials evaluating prospectively their potential in adults with cancer but none in children so far.

The Objective is to determine the Maximal Tolerated Dose (MTD) of a combination of oral metronomic vinorelbine and daily oral propranolol. This study is a phase I trial with a "rolling six" design and a dose escalation with thrice weekly oral vinorelbine only plus addition of daily oral propranolol after completion of the first cycle. PK analysis of vinorelbine and propranolol will be performed. Once the recommended dose of the combination established 4 extension cohorts of 9 patients will be added Potential biomarkers (such as beta-adrenergic receptors on the tumours, B-tubulin isotypes in the tumour) will also be evaluated.

This will provide a well tolerated, all oral combination for patients with refractory/relapsing tumours. This combination could also be then proposed as a maintenance for instance in patients with rhabdomyosarcoma or neuroblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant solid tumour and refractory low grade gliomas and desmoids tumours.
* Relapsed or refractory tumours after at least one line of treatment (patients can have been previously treated with oral or IV vinorelbine with a weekly schedule)
* Measurable targets
* Lansky Score > 70 or score OMS < 2.
* Life expectancy > 6 months.
* Adequate haematological function: neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 75 x 109/L
* Creatinine< 1.5X normal value for the age or clearance >70 ml/mn/1.73 m2
* Liver function: Bilirubin < 3N and ALAT and ASAT < 4 N).
* Other organ toxicity < Grade 2 according to NCI-CTC version 4.0
* No active infection

Exclusion Criteria:

* Absence of a wash out period of:

  * 21 days in case of previous chemotherapy or targeted therapy (reduced to 2 weeks in case of treatment vincristine or prolonged to 6 weeks in case of treatment with nitrosurea agents)
  * 6 weeks in case of prior radiotherapy of the target lesions
* Peripheral neuropathy > grade 2
* contra-indication to Propranolol (i.e. asthma, bradycardia, hypotension, decreased SF, ECG-anomalies)
* Pregnancy or breast feeding

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
number of patients with grade 3 toxicity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France